CLINICAL TRIAL: NCT05158907
Title: Patient Reported Scale vs CTCAE Grading for Reporting Chemotherapy Related Adverse Effects: A Prospective Comparator Study
Brief Title: Patient Reported Scale vs CTCAE Grading: A Prospective Comparator Study
Acronym: PROSE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient recruitment is slow
Sponsor: Tata Medical Center (Other)
Responsible Party: Principal Investigator, Tanuj Chawla, Principal Investigator, Tata Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2021/TMC/239/IRB50
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient reported adverse event scale will be given to study participants
Who Masked: Care Provider, Investigator
Masking Description: The clinician will not get the opportunity to see the patient reported scale until the end of patient's participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient reported Adverse event scale — Participants will be given a patient reported AE scale with numbers from 0 to 10 before start of each chemotherapy cycle. The PRAE scale will be like a Visual Analogue Scale and the patients will be given instructions how to record AEs that they experience after each chemotherapy cycle, until the first radiological assessment is done (palliative settings) or after 4 cycles of chemotherapy in adjuvant settings. Participants will take scale home to record the adverse effects and give it a number. Only the most severe will be analyzed. When patient reports for the next cycle of chemotherapy they will be asked to deposit the scale before meeting the physician. The physician will ask patient about the AEs experienced with the chemotherapy and record them using CTCAE grade. The study participants, at the start of chemotherapy cycle, will be informed, as a standard practice, to report to the emergency or contact nearest local clinic/hospital if the AE is severe or can't be managed at home.

SUMMARY:
Over a million new cancer cases are diagnosed in India each year. This huge burden coupled with inadequate infrastructural facilities is adversely affecting the quality of patient care. As a side effect it is adding to cost of health care which patient is paying from his/her own pocket. Total care of cancer patients taking chemotherapy is interrupted by several obstacles some of which can be prevented or detected early and treated. Most of the patients experience toxicity during cancer chemotherapy but the reporting remains inadequate as patients are not aware how to report or the physicians, many a times, are extremely busy to record and act on them early. We assume that using patient reported adverse event (AE) scale is more practical and easier to use for reporting AEs. This intervention, we feel, can pick more AEs which can lead to early intervention by the physician and ultimately reducing the cost of treatment to patients. We plan to include adult patients (>18years) having Gastro-intestinal cancers (both colorectal and non-colorectal cancers) who are scheduled to receive combination chemotherapy medicines with both curative and non-curative intent (in patients with advanced cancers). Patients will be given an AE scale and will be asked to fill it at home during each chemotherapy cycle, for upto 4 cycles. The physician will also ask them about the AE during the next clinic visit and record the AEs as per the widely accepted AE scale (Common Terminology Criteria for Adverse Events-CTCAE) for reporting. The patient reported AE scale will then be compared and analyzed with standard CTCAE using relevant statistical methods.

DETAILED DESCRIPTION:
Population and setting: This study will be conducted at Tata Medical Center (TMC), Kolkata. Patients in TMC are managed using evidence-based treatment protocols and through multidisciplinary teams. Patients in this study will be drawn from those attending the cancer clinics. Adult patients (>18years age) receiving combination anti-cancer chemotherapy for gastro-intestinal cancers (colorectal and non-colorectal) will be enrolled.

Trial design: This is a single centre prospective study. Patients who provide written consent for the study will be enrolled. Most commonly used standard combination chemotherapy regimens used in our clinic will be taken in this study i.e., weekly (e.g., Paclitaxel-Carboplatin, Gemcitabine-Cisplatin), biweekly (e.g. FOLFOX/FOLFIRI/ FOLFOXIRI/FLOT/DCF/GEMOX), once every three weeks (e.g. Capox/CapIri/mDCF) or once every 4 weeks (e.g. ETOCIS/Capecitabine-Temozolomide) with or without Targeted therapy (e.g. Bevacizumab/Cetuximab/Panitumumab) and/or Immunotherapy (e.g. Pembrolizumab/ Nivolumab/Atezolizumab/Ipilimumab). No single agent chemotherapy will be considered. Patients will be stratified to type of combination chemotherapy with high and low probability of causing severe toxicities. This will be based on our experience in clinical practice. Chemotherapy combinations with high probability are FOLFOXIRI, FLOT, Capiri (Xeliri), mDCF and with low probability are FOLFOX, FOLFIRI, GEMOX, Gemcitabine-Cisplatin, Paclitaxel-Carboplatin, CapOx, ETOCIS, Capecitabine-Temozolomide.

Intervention: Consenting patients will be given a patient reported AE (PRAE) scale with numbers from 0 (Nil) to 10 (most severe) before start of each chemotherapy cycle. This AE scale will have pre-defined symptom related AEs with the provision of adding some more by the patient if they have those symptoms. The PRAE scale will be like a Visual Analogue Scale (VAS) and the patients will be given instructions how to record AEs that they experience after each chemotherapy cycle, until the first radiological assessment is done (palliative settings) or after 4 cycles of chemotherapy in adjuvant settings. They will be asked to take the scale home to record the adverse effects and give it a number (as per VAS), depending on the severity. They will be told to record all the AEs (whenever they experience), even if same AE happens more than once during a particular chemotherapy. Only the most severe one will be analysed. When patient reports for the next cycle of chemotherapy he/she will be asked to deposit the PRAE scale with the study co-ordinator before meeting the treating physician and a new copy of a blank scale will be given to him/her for the next cycle. In the clinic, as a standard practice, the doctor will ask the patient about the AEs experienced with the previous chemotherapy and record them as per the CTCAE, grade, version 5. The clinician will not get the opportunity to see the patient reported scale until the end of patient's participation in the study. All the study participants, at the start of chemotherapy and before each chemotherapy cycle, will be informed, as a standard practice, to report to the emergency or contact nearest local clinic/hospital if the AE is severe or can't be managed at home. The response by patients will be analysed for the pre-defined outcomes. The management of side effects is beyond the scope of this study and will be managed as per the standard clinical practice in TMC. The cost of which will be borne by the patient or his/her insurance company.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with more than 18years of age.
* Provide written informed consent
* Diagnosed with Gastrointestinal cancer (both colorectal and non-colorectal cancer of all histological types) and are planned for adjuvant or palliative combination chemotherapy with or without Targeted therapy and Immunotherapy.
* Patients who have been fully recovered from cancer surgery, if any.
* Residing within 50km radius of TMC.
* Patient or their family member who can read, write and comprehend Bangla, Hindi or English language.

Exclusion Criteria:

* Patients not residing in India e.g. patients from neighbouring countries like Bangladesh, Nepal, Bhutan.
* Patients whose comorbid conditions like diabetes, hypertension, hypo/hyperthyroidism, heart ailment are not under control.
* Patient who is not willing to start or continue the medicines for their comorbid conditions.
* Patients with psychomotor comorbid conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement in detection rate of adverse effects of patient reported adverse effect (AE) scale versus the standard CTCAE grading by a physician. | 1 year
  Proposed AE scale will be compared with standard CTCAE scale

SECONDARY OUTCOMES:
Patient Compliance to filling the patient reported AE scale. | 1 year
  Will see how many patients will be able to fill the new scale
Early intervention using patient reported AE scale and preventing severity of AE in the subsequent chemotherapy cycles. | 1 year
  Whether AE scale can prevent severity of adverse events
Timely chemotherapy dose adjustments using patient reported adverse effect scale | 1 year
  Chemotherapy doses can be adjusted if early adverse effects can be picked using AE scale.
Reduction in cost of cancer care using patient reported AE scale. | 1 year
  Whether cost of cancer can be reduced using the proposed scale

CONTACTS AND LOCATIONS:
Overall Officials: Tanuj Chawla, MD, Principal Investigator — Tata Medical Center
Locations (1):
- Tata Medical Center, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No